CLINICAL TRIAL: NCT02936882
Title: Evaluation of Antral Ultrasonography for Full Stomach Diagnosis Before Pediatric Surgical Emergencies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Olivier MAUPAIN, Medical Doctor, Hôpital Necker-Enfants Malades
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DAR_NCK_OMN0001
Record Dates: First submitted 2016-10-06; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Content; Full Stomach Status
Keywords: ultrasonography; aspiration; emergency; children; antrum
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative gastric ultrasonography (Other)
  Interventions: Procedure: Preoperative gastric ultrasonography

INTERVENTIONS:
Procedure: Preoperative gastric ultrasonography — Before surgical emergency procedure, a preoperative antral ultrasonography is performed to assess gastric content.

SUMMARY:
This study evaluates antral ultrasonography for the diagnosis of full stomach before surgical emergencies in pediatric population. Preoperative ultrasonographic antral evaluation is compared to peroperative gastric aspirate with nasogastric tube.

ELIGIBILITY:
Inclusion Criteria:

* Surgical emergency procedure
* ASA I-II

Exclusion Criteria:

* Ultrasound antrum assessment not possible
* No nasogastric tube during surgery
* Vital emergency
* Patient from Critical Care Ward
* Time between ultrasound assessment and gastric content collecting up to 20min
* Child and/or Parents doesn't/don't want to participate in the study
* Personal medical history of gastric or oesophagus desease

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Volume of gastric content aspirated throw nasogastric tube | 20 min

SECONDARY OUTCOMES:
Grades as described by Perlas et al. for ultrasonographic qualitative evaluation of gastric content | 20 min
relationship between peroperative gastric content and ultrasonographic antrum assessment | 20 min
Time to perform antral ultrasonography | 20 min
Quality of image obtained during antral ultrasonography | 20 min
Child behaviour during antral ultrasonography | 20 min
Number of participants with exploitable antral ultrasonography | 20 min
Reasons for antral ultrasonography failure | 20 min

CONTACTS AND LOCATIONS:
Locations (1):
- Necker Enfants-Malades University Hospital - APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided